CLINICAL TRIAL: NCT05238220
Title: Utilization of the Viracor® Assay in Directing Duration of Valganciclovir Prophylaxis in CMV High Risk Kidney Transplant Recipients
Brief Title: Utilization of the Viracor® Assay for Valganciclovir Prophylaxis in CMV High Risk Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Piedmont Healthcare (Other)
Collaborators: ViraCor Laboratories (Industry)
Responsible Party: Principal Investigator, Christina Klein, Transplant Nephrologist, Piedmont Healthcare
Other Study IDs: Viracor
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — Valganciclovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- continue valganciclovir prophylaxis: continue valganciclovir prophylaxis for up to 12 months total when anti-CMV immunity absent
  Interventions: Drug: Valganciclovir
- discontinue valganciclovir prophylaxis: discontinue valganciclovir prophylaxis when anti-CMV immunity present after routine care prophylaxis

INTERVENTIONS:
Drug: Valganciclovir — continuation of valganciclovir prophylaxis up to 12 months with absence of demonstrated anti-CMV immunity
  Groups: continue valganciclovir prophylaxis

SUMMARY:
The purpose of this study is to evaluate whether the use of the Viracor® CMV immunity assay at 6 months post-transplant in CMV high risk kidney transplant recipients would help identify those patients at higher risk of post-prophylaxis CMV viremia or disease and thereby select those patients in which a longer duration of valganciclovir prophylaxis would be beneficial.

DETAILED DESCRIPTION:
Kidney transplant patients that are cytomegalovirus (CMV) seronegative (IgG negative) at time of transplant and receive a graft from a donor that is CMV seropositive (IgG positive) are at increased risk of developing post-transplant CMV viremia and disease. These patients receive standard CMV prophylaxis with valganciclovir for 6 months post-transplant. However, a considerable proportion of these patients (25 - 42% at our center over the last 5 years) will go on to develop CMV viremia and/or disease after this valganciclovir prophylaxis is discontinued. To date, there is no strong data regarding whether certain patients would benefit from extension of valganciclovir prophylaxis beyond the standard 6-month period.

The purpose of this study is to evaluate whether the use of the Viracor® CMV immunity assay at 6 months post-transplant in CMV high risk kidney transplant recipients would help identify those patients at higher risk of post-prophylaxis CMV viremia or disease and thereby select those patients in which a longer duration of valganciclovir prophylaxis would be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent
* Kidney Transplant Recipients
* Classified as CMV high risk at time of transplant (donor CMV IgG positive and recipient CMV IgG negative)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CMV High Risk Kidney Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Use of Viracor CMV immunity assay | 6 months post-transplant through 12 months prophylaxis
  continue valganciclovir prophylaxis for additional time due to absence of demonstrated anti-CMV immunity

CONTACTS AND LOCATIONS:
Locations (1):
- Piedmont Atlanta Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No